CLINICAL TRIAL: NCT03296787
Title: A Phase 1, Open-Label, Parallel Group Trial to Evaluate the Effect of Renal Impairment and Dialysis Treatment on the Pharmacokinetics of a Single Intravenous Dose of TAK-954
Brief Title: A Study to Evaluate the Effect of Renal Impairment and Dialysis Treatment on the Pharmacokinetics (PK) of a Single Intravenous (IV) TAK-954
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-954-1007; U1111-1196-9206 (Registry Identifier: WHO); 2017-000715-16 (EudraCT Number)
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Renal Impairment; Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A TAK-954 0.2 mg: Healthy Participants (Experimental): Participants with normal renal function receive TAK-954 0.2 milligram (mg), infusion, intravenously in fasted state, once on Day 1 of a 6-day period.
  Interventions: Drug: TAK-954
- Group B TAK-954 0.2 mg: Mild Renal Impairment (Experimental): Participants receive TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period.
  Interventions: Drug: TAK-954
- Group C TAK-954 0.2 mg: Moderate Renal Impairment (Experimental): Participants receive TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period.
  Interventions: Drug: TAK-954
- Group D TAK-954 0.2 mg: Severe Renal Impairment (Experimental): Participants without hemodialysis or End-stage Renal Disease (ESRD) receive TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period.
  Interventions: Drug: TAK-954
- Group E TAK-954 0.2 mg: End-stage Renal Disease (ESRD) (Experimental): Participants with hemodialysis receive TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 4-day period followed by a minimum 13-day washout period, further followed by TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 4-day period.
  Interventions: Drug: TAK-954

INTERVENTIONS:
Drug: TAK-954 — TAK-954 intravenous infusion.

SUMMARY:
The purpose of this study is to evaluate the effect of varying degrees of renal function on the PK of TAK-954 following single-dose IV administration and to investigate the impact of hemodialysis on the PK of single IV doses of TAK-954.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. This study will evaluate the effect of varying degrees of renal function on the PK of TAK-954 following single-dose IV administration and to investigate the impact of hemodialysis on the PK of single IV doses of TAK-954.

The study will enroll approximately up to 40 participants. Participants will be enrolled in one of the 5 treatment groups based on their renal impairment which will be determined based on Cockcroft and Gault (CG) equation as follows:

* Group A TAK-954 0.2 mg: Healthy Participants
* Group B TAK-954 0.2 mg: Mild Renal Impairment
* Group C TAK-954 0.2 mg: Moderate Renal Impairment
* Group D TAK-954 0.2 mg: Severe Renal Impairment or End-stage Renal Disease (ESRD) Without Hemodialysis
* Group E TAK-954 0.2 mg: End-stage Renal Disease (ESRD) With Hemodialysis

All participants in groups A to D will receive a single dose of TAK-954 and two single doses in Group E.

Enrollment in Group B (Mild) and Group E (ESRD requiring dialysis) will be based on assessment of safety and available PK data from Group C and Group D respectively.

This multi-center trial will be conducted in Czech Republic and Hungary. The overall time to participate in this study is approximately 8 weeks. Participants in Groups A to D will remain confined to clinic for 3 days. For both treatments, participants in Group E requiring dialysis will remain confined to clinic for 3 days. All participants will make a final visit to the clinic 10-14 days after receiving their last dose for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. All participants: Male and female participants (non-childbearing potential) who are aged 18 to 75 years, inclusive, with a body mass index (BMI) between 18 to 35 kilogram per square meter (kg/m^2).
2. Group A: As much as possible, the healthy participants with normal renal function (creatinine clearance [CLcr] greater than or equal to [>=] 90 milliliter per minute [mL/min]) should be comparable to participants with renal impairment with respect to median age and weight (approximately 50 percent [%] of healthy participants on each side of the median age and weight of currently enrolled renally-impaired participants grouped together), sex, and race. This will be decided by the investigators in discussion with Takeda.
3. Groups B to E: Participants who have stable RI, defined as no clinically significant change in disease status, as documented by the participant's most recent CLcr assessment; serum creatinine must not vary more than approximately 30% from Screening to Day -1 to confirm stable disease. Participants should also be in good health commensurate with their renal status.

   * Group B: Participants with mild RI (CLcr 60 to less than [<] 90 mL/min).
   * Group C: Participants with moderate RI (CLcr 30 to <60 mL/min).
   * Group D: Participants with severe RI or ESRD but not requiring dialysis (CLcr <30 mL/min).
   * Group E: Participants with ESRD requiring dialysis (<15 mL/min requiring hemodialysis at least 3 times/week, and having been on the same dialysis treatment regimen for at least 1 month before trial entry).
4. Participants should be on a stable drug regimen defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) before dosing with TAK-954.

Exclusion Criteria:

1. All participants:

   * Are renal allograft recipients within 1 year of screening.
   * Have a history of gastrointestinal (GI) motility disorder or intestinal obstruction.
   * Have urinary incontinence without catheterization.
2. Group A: Participants who, in the discretion of the investigator, have a history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases will be excluded from the trial.
3. Groups B to E:

   * Receive dialysis other than intermittent dialysis (except Group E).
   * Have renal disease secondary to hepatic disease (hepatorenal syndrome).
   * At the discretion of the investigators, have any significant hepatic, cardiac, or pulmonary disease or participants who are clinically nephrotic.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- Czechia (2):
  - PRA CZ, s.r.o, Prague, Prague
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
- Hungary (2):
  - PRA Magyarorszag Kft., Budapest
  - Szent Imre Egyetemi Oktatokorhaz Belgyogyazati Szakmak Matrix Intezet, Budapest

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Czech Republic and Hungary from 21 November 2017 to 09 August 2019.
Pre-assignment Details: Participants with normal renal function and renal impairment were enrolled in 1 of the 4 groups: A (healthy), C (moderate), D (severe), and E (end-stage renal disease [ESRD]) to receive TAK-954 0.2 milligram (mg). Based on available safety and pharmacokinetics (PK) data from Group C, participants were not enrolled in Group B (mild).
Groups:
- Group A: Healthy Participants: TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period (Treatment 1), followed by a minimum 13-day washout period, further followed by probe cocktail of different cytochrome P-450 (CYP) substrates (caffeine 100 mg, oral [CYP1A2] + midazolam 0.025 milligram per kilogram [mg/kg], intravenously [CYP3A4]), once on Day 1 of a 4-day period (Treatment 2) in participants with normal renal function.
- Group C: Moderate Renal Impairment: TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period (Treatment 1), followed by a minimum 13-day washout period, further followed by probe cocktail of different CYP substrates (caffeine 100 mg, oral [CYP1A2] + midazolam 0.025 mg/kg, intravenously [CYP3A4]), once on Day 1 of a 4-day period (Treatment 2) in participants with moderate renal impairment.
- Group D: Severe Renal Impairment Not Requiring Dialysis: TAK-954 0.2 mg, infusion, intravenously in fasted state, once on Day 1 of a 6-day period (Treatment 1) in participants with severe renal impairment or ESRD without dialysis.
- Group E: ESRD Requiring Dialysis: TAK-954 0.2 mg, infusion, intravenously in fasted state, 1 hour after the end of dialysis, once on Day 1 of a 6-day Period 1, followed by a minimum 13-day washout period, further followed by TAK-954 0.2 mg, infusion, intravenously in fasted state, 2 hours before the start of dialysis, once on Day 1 of a 4-day Period 2 in participants with ESRD requiring dialysis.
Period: Overall Study
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis | Group E: ESRD Requiring Dialysis
Started | 8 | 8 | 9 | 7
Completed | 8 | 8 | 9 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who were enrolled and received at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis | Group E: ESRD Requiring Dialysis | Total
Number analyzed (Participants) | 8 | 8 | 9 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (15.62) | 70.6 (3.50) | 62.2 (11.03) | 52.6 (10.06) | 60.9 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 0 | 11
  Male | 5 | 4 | 5 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 9 | 7 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 9 | 7 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 6 | 6 | 5 | 3 | 20
  Hungary | 2 | 2 | 4 | 4 | 12
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 79.95 (7.773) | 75.95 (13.035) | 76.22 (14.457) | 82.39 (7.006) | 78.43 (11.072)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.88 (4.051) | 26.25 (4.166) | 27.33 (4.272) | 28.14 (2.673) | 27.13 (3.765)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.25 (9.706) | 170.25 (9.543) | 166.89 (9.519) | 171.00 (6.976) | 170.22 (8.965)
Creatine Clearance [Mean (Standard Deviation); unit: milliliter per minute (mL/min)] | 107.11 (23.417) | 46.20 (10.767) | 23.20 (6.385) | 10.54 (2.504) | 47.16 (39.484)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliter per minute/1.73 square meter] | 89.93 (13.779) | 41.68 (11.527) | 18.13 (8.648) | 6.93 (2.757) | 39.52 (33.514)

OUTCOME MEASURES:

1. Primary Outcome: Groups A, C and D; Cmax: Maximum Observed Plasma Concentration for TAK-954 (Total and Free)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 120 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received at least 1 dose of trial drug and had at least 1 measurable TAK-954 plasma concentration. The outcome measure (OM) was planned to be assessed for the groups where blood samples were collected before the start of TAK-954 infusion and through 120 hours post-infusion.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter (ng/mL)
  TAK-954 (Total) | 2.623 (12.8) | 2.536 (23.2) | 2.660 (17.6)
  TAK-954 (Free) | 0.1270 (29.2) | 0.1282 (22.5) | 0.1572 (21.7)
Statistical Analysis 1: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Total): An analysis of variance (ANOVA) were performed on log transformed Cmax (total TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.7265, ANOVA
Statistical Analysis 2: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed Cmax (total TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.9839, ANOVA
Statistical Analysis 3: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of Cmax (free TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.9393, ANOVA
Statistical Analysis 4: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of Cmax (free TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.1321, ANOVA

2. Primary Outcome: Groups A, C and D; AUC(0-72): Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Post-dose for TAK-954 (Free and Total)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 72 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received at least 1 dose of trial drug and had at least 1 measurable TAK-954 plasma concentration. The OM was planned to be assessed for the groups where blood samples were collected before the start of TAK-954 infusion and through 120 hours post-infusion.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
hour*nanogram per milliliter (h*ng/mL)
  TAK-954 (Total) | 22.25 (19.1) | 24.91 (22.9) | 28.62 (18.1)
  TAK-954 (Free) | 1.078 (25.7) | 1.259 (25.1) | 1.690 (25.9)
Statistical Analysis 1: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUC(0-72) (total TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.3600, ANOVA
Statistical Analysis 2: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUC(0-72) (total TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0816, ANOVA
Statistical Analysis 3: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUC(0-72) (free TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.2686, ANOVA
Statistical Analysis 4: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUC(0-72) (free TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0059, ANOVA

3. Primary Outcome: Groups A, C and D; AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-954 (Free and Total)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 120 hours) post-infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL
  TAK-954 (Total) | 24.39 (17.7) | 30.00 (20.0) | 34.28 (19.3)
  TAK-954 (Free) | 1.184 (26.8) | 1.516 (24.3) | 2.025 (26.7)
Statistical Analysis 1: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUClast (total TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.0998, ANOVA
Statistical Analysis 2: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUClast (total TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0155, ANOVA
Statistical Analysis 3: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUClast (free TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.0916, ANOVA
Statistical Analysis 4: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUClast (free TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0014, ANOVA

4. Primary Outcome: Groups A, C and D; AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-954 (Free and Total)
Time Frame: Day 1 pre-infusion and at multiple time points (up to 120 hours) post-infusion
Population: PK set:participants who enrolled and received at least 1 dose of trial drug and had at least 1 measurable TAK-954 plasma concentration. Here,"overall number of participants analyzed": participants who were evaluable for this OM. OM was planned to be assessed in groups where blood samples collected pre-TAK-954 infusion up to 120 hours post-infusion.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 7 | 7
h*ng/mL
  TAK-954 (Total) | 25.43 (16.8) | 34.90 (16.2) | 38.59 (23.9)
  TAK-954 (Free) | 1.234 (28.4) | 1.749 (24.8) | 2.320 (29.7)
Statistical Analysis 1: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUC∞ (total TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.0038, ANOVA
Statistical Analysis 2: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Total): An ANOVA were performed on log transformed AUC∞ (total TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0004, ANOVA
Statistical Analysis 3: Comparison: Group A: Healthy Participants vs Group C: Moderate Renal Impairment; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUC∞ (free TAK-954) to compare moderate renal impairment group with the normal renal function group; p = 0.0389, ANOVA
Statistical Analysis 4: Comparison: Group A: Healthy Participants vs Group D: Severe Renal Impairment Not Requiring Dialysis; Test type: Superiority — TAK-954 (Free): An ANOVA were performed on natural logarithm of AUC∞ (free TAK-954) to compare severe renal impairment group with the normal renal function group; p = 0.0011, ANOVA

5. Primary Outcome: Groups A, C and D; Ae: Amount of TAK-954 Excreted in Urine
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received at least 1 dose of trial drug and had at least 1 measurable TAK-954 plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
milligram (mg) | 0.03797 (0.011633) | 0.01763 (0.0087713) | 0.01190 (0.0091124)

6. Primary Outcome: Group E; Ae: Amount of TAK-954 Excreted in Urine in Period 1
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received at least 1 dose of trial drug and had at least 1 measurable TAK-954 plasma concentration. Here, "overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: mg
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 5
mg | 0.0003489 (0.00021788)

7. Primary Outcome: Group E; Ae: Amount of TAK-954 Excreted in Urine in Period 2
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: mg
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 4
mg | 0.001240 (0.00062000)

8. Primary Outcome: Groups A, C and D; Fe: Fraction of TAK-954 Excreted in Urine
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: percentage of TAK-954 dose
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
percentage of TAK-954 dose | 19.00 (5.8075) | 8.808 (4.3746) | 5.953 (4.5595)

9. Primary Outcome: Group E; Fe: Fraction of TAK-954 Excreted in Urine in Period 1
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: percentage of TAK-954 dose
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 5
percentage of TAK-954 dose | 0.1739 (0.10869)

10. Primary Outcome: Group E; Fe: Fraction of TAK-954 Excreted in Urine in Period 2
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: percentage of TAK-954 dose
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 4
percentage of TAK-954 dose | 0.6190 (0.30950)

11. Primary Outcome: Groups A, C and D; CLR: Renal Clearance for TAK-954
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: The PK set consisted of all participants who were enrolled and received at least 1 dose of study drug and had at least 1 measurable TAK-954 plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis
Number analyzed (Participants) | 8 | 8 | 8
liter per hour (L/h) | 2.629 (0.78762) | 1.255 (0.51478) | 0.6836 (0.56141)

12. Primary Outcome: Group E; CLR: Renal Clearance for TAK-954 in Period 1
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 5
L/h | 0.03192 (0.017670)

13. Primary Outcome: Group E; CLR: Renal Clearance for TAK-954 in Period 2
Time Frame: Day 1 pre-infusion and at multiple time points (up to 24 hours) post-infusion
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 4
L/h | 0.08330 (0.041650)

14. Primary Outcome: Group E; CLD: Clearance of Dialysate for TAK-954 in Period 2
Time Frame: Day 1 pre-infusion and at multiple time points (up to 4 hours) post-infusion
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group E: ESRD Requiring Dialysis
Number analyzed (Participants) | 7
L/h | 1.368 (30.0)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug and no more than 14 days after the last dose of study drug as Treatment 2 (up to Day 29) in Group A, C, and E), and Treatment 1 (up to Day 15) in for Group D
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. TEAEs includes adverse events occurred during Treatments 1 and 2 in Groups A and C, as planned.
Groups:
- Group E: ESRD 1 Hour After Dialysis: TAK-954 0.2 mg, infusion, intravenously in fasted state, 1 hour after the end of dialysis, once on Day 1 of a 6-day Period 1 in participants with ESRD requiring dialysis.
- Group E: ESRD 2 Hours Before Dialysis: TAK-954 0.2 mg, infusion, intravenously in fasted state, 2 hours before the start of dialysis, once on Day 1 of a 4-day Period 2 in participants with ESRD requiring dialysis.
Arm/Group | Group A: Healthy Participants | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment Not Requiring Dialysis | Group E: ESRD 1 Hour After Dialysis | Group E: ESRD 2 Hours Before Dialysis
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 2/9 | 1/7 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Healthy Participants (N=8) | Group C: Moderate Renal Impairment (N=8) | Group D: Severe Renal Impairment Not Requiring Dialysis (N=9) | Group E: ESRD 1 Hour After Dialysis (N=7) | Group E: ESRD 2 Hours Before Dialysis (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03296787/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03296787/SAP_001.pdf